CLINICAL TRIAL: NCT05343598
Title: Empirical Validation of a Cerebellar-cortical Hallucination Circuit
Brief Title: Using Transcranial Magnetic Stimulation (TMS) to Understand Hallucinations in Schizophrenia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Mark A. Halko, PhD, Assistant Professor of Psychiatry, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2021P002459; R01MH126000 (NIH)
Record Dates: First submitted 2022-04-13; First posted 2022-04-25 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Schizophrenia; Schizo Affective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The subjects, care providers, investigators and outcome assessors will all be blinded as to the randomization sequence, and thus will be blinded as to sham vs active TMS status. Blinding codes are used to determine which side of an active/passive Magpro coil (cool B65 A/P, Magventure A/S, Denmark) is used for stimulation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active cerebellum rTMS (Active Comparator): Cerebellar targeted iTBS, twice daily, one week.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)
- Sham cerebellum rTMS (Sham Comparator): Cerebellar targeted sham iTBS, twice daily, one week.
  Interventions: Device: Sham Repetitive Transcranial Magnetic Stimulation (rTMS)

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — rTMS is a technique of TMS that allows for selective external manipulation of neural activity in a non-invasive manner. During rTMS a rapidly changing current is passed through an insulated coil placed against the scalp. This generates a temporary magnetic field, which in turn induces electrical current in neurons and allows for modulation of neural circuitry.
  The rTMS pulses will be delivered in a pattern consisting of 2 s trains of 3 pulses at 50 Hz, repeated at 5 Hz every 10s for 600 total pulses.
  Other Names: iTBS
  Arms: Active cerebellum rTMS
Device: Sham Repetitive Transcranial Magnetic Stimulation (rTMS) — rTMS is a technique of TMS that allows for selective external manipulation of neural activity in a non-invasive manner. During rTMS a rapidly changing current is passed through an insulated coil placed against the scalp. This generates a temporary magnetic field, which in turn induces electrical current in neurons and allows for modulation of neural circuitry.
  The rTMS pulses will be delivered in a pattern consisting of 2 s trains of 3 pulses at 50 Hz, repeated at 5 Hz every 10s for 600 total pulses.
  Sham is achieved by using a coil with a magnetic shield preventing magnetic field from reaching the head.
  Other Names: iTBS
  Arms: Sham cerebellum rTMS

SUMMARY:
This study uses a noninvasive technique called transcranial magnetic stimulation (TMS) to study how hallucinations work in schizophrenia.

TMS is a noninvasive way of stimulating the brain, using a magnetic field to change activity in the brain. The magnetic field is produced by a coil that is held next to the scalp. In this study the investigators will be stimulating the brain to learn more about how TMS might improve these symptoms of schizophrenia.

DETAILED DESCRIPTION:
This study tests the hypothesis that hallucinations in schizophrenia are mediated by network pathophysiology, and that network pathophysiology can be quantified by the functional connectivity of a cerebellar-thalamo-cortical circuit. To accomplish this, participants will be recruited who are diagnosed with schizophrenia or schizoaffective disorder who experience auditory hallucinations.

Participants will undergo an initial screening session to complete informed consent and undergo baseline assessments of schizophrenia symptom severity. These assessments include reporter-based measures such as the Positive and Negative Syndrome Scale (PANSS).

Participants will then undergo an MRI scan that includes structural and resting-state functional magnetic resonance imaging (rsfMRI). These rsfMRI imagines will be used to isolate individual resting state networks for targeting of rTMS modulation.

Participants will then undergo five days of twice daily rTMS sessions.

One week after the last rTMS session, participants will undergo follow-up MRI imaging and the same study assessments.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia or schizoaffective disorder

Exclusion Criteria:

* substance use disorder in past 3 months
* ambidexterity
* contraindications for TMS or MRI including :
* history of neurological disorder
* history of head trauma resulting in loss of consciousness
* history of seizures or diagnosis of epilepsy or first degree relative family history of epilepsy
* metal in brain or skull
* implanted devices such as a pacemaker, medication pump, nerve stimulator or ventriculoperitoneal shunt
* claustrophobic in MRI

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2021-10-13 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
functional connectivity | baseline, 1 week after TMS
  change in functional connectivity of a putative cerebellar-thalamic-cortical hallucination circuit (cerebellum to thalamus) will be assessed before and after (1 week followup) TMS stimulation.
Positive and Negative Syndrome Scale (PANSS) | baseline
  The PANSS is clinical rating scale of symptom severity . Each descriptor is rated on a 7 point scale from 1=(absence of any symptom) to 7=(extremely severe symptoms).
Scale for the Assessment of Positive Symptoms (SAPS) | baseline
  The SAPS is clinical rating scale of symptom severity . Each descriptor is rated on a 5 point scale from 1=(absence of any symptom) to 5=(extremely severe symptoms).
Auditory Hallucination Rating Scale (AHRS) Scale (AHRS) | baseline
  The AHRS is a 7-item clinical rating scale used to assess auditory hallucinations.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Halko, PhD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
deidentified participant data will be shared with NIMH Data Repository (NDA).

REFERENCES:
- [Background] Brady RO Jr, Gonsalvez I, Lee I, Ongur D, Seidman LJ, Schmahmann JD, Eack SM, Keshavan MS, Pascual-Leone A, Halko MA. Cerebellar-Prefrontal Network Connectivity and Negative Symptoms in Schizophrenia. Am J Psychiatry. 2019 Jul 1;176(7):512-520. doi: 10.1176/appi.ajp.2018.18040429. Epub 2019 Jan 30. PMID 30696271
- [Background] Basavaraju R, Ithal D, Thanki MV, Ramalingaiah AH, Thirthalli J, Reddy RP, Brady RO Jr, Halko MA, Bolo NR, Keshavan MS, Pascual-Leone A, Mehta UM, Kesavan M. Intermittent theta burst stimulation of cerebellar vermis enhances fronto-cerebellar resting state functional connectivity in schizophrenia with predominant negative symptoms: A randomized controlled trial. Schizophr Res. 2021 Dec;238:108-120. doi: 10.1016/j.schres.2021.10.005. Epub 2021 Oct 12. PMID 34653740
- [Background] Nawaz U, Lee I, Beermann A, Eack S, Keshavan M, Brady R. Individual Variation in Functional Brain Network Topography is Linked to Schizophrenia Symptomatology. Schizophr Bull. 2021 Jan 23;47(1):180-188. doi: 10.1093/schbul/sbaa088. PMID 32648915
- [Background] Hwang M, Roh YS, Talero J, Cohen BM, Baker JT, Brady RO, Ongur D, Shinn AK. Auditory hallucinations across the psychosis spectrum: Evidence of dysconnectivity involving cerebellar and temporal lobe regions. Neuroimage Clin. 2021;32:102893. doi: 10.1016/j.nicl.2021.102893. Epub 2021 Nov 24. PMID 34911197
- [Background] Brady RO Jr, Beermann A, Nye M, Eack SM, Mesholam-Gately R, Keshavan MS, Lewandowski KE. Cerebellar-Cortical Connectivity Is Linked to Social Cognition Trans-Diagnostically. Front Psychiatry. 2020 Nov 4;11:573002. doi: 10.3389/fpsyt.2020.573002. eCollection 2020. PMID 33329111
- [Background] Ward HB, Brady RO Jr, Halko MA. Bridging the Gap: Strategies to Make Psychiatric Neuroimaging Clinically Relevant. Harv Rev Psychiatry. 2021 May-Jun 01;29(3):185-187. doi: 10.1097/HRP.0000000000000295. PMID 33882534
- [Background] Halko MA, Farzan F, Eldaief MC, Schmahmann JD, Pascual-Leone A. Intermittent theta-burst stimulation of the lateral cerebellum increases functional connectivity of the default network. J Neurosci. 2014 Sep 3;34(36):12049-56. doi: 10.1523/JNEUROSCI.1776-14.2014. PMID 25186750
- [Background] Huang YZ, Edwards MJ, Rounis E, Bhatia KP, Rothwell JC. Theta burst stimulation of the human motor cortex. Neuron. 2005 Jan 20;45(2):201-6. doi: 10.1016/j.neuron.2004.12.033. PMID 15664172